CLINICAL TRIAL: NCT01567241
Title: Prospective Off-center Randomised Trial of Clinical Hypnosis Versus Relaxation Music
Brief Title: Clinical Hypnosis During Insemination or Embryotransfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, PD Dr. med. Joscha Reinhard, MBBS BSc(Hon), Principal investigator, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 329/11
Record Dates: First submitted 2012-03-22; First posted 2012-03-30 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Reproduction Dysfunction
Keywords: clinical hypnosis; relaxation music; reproduction techniques; insemination; embryo transfer; pregnancy rate
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation music (Placebo Comparator)
  Interventions: Other: clinical hypnosis or relaxation music
- Clinical hypnosis (Experimental)
  Interventions: Other: clinical hypnosis or relaxation music

INTERVENTIONS:
Other: clinical hypnosis or relaxation music — 25 minute tape recording

SUMMARY:
Does clinical hypnosis or relaxation music improve the pregnancy rate if reproduction techniques are required?

ELIGIBILITY:
Inclusion Criteria:

Planned insemination or embryo transfer

Exclusion Criteria:

under age not able to understand German

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 4 weeks after insemination / embryotransfer
  Outpatient follow up after insemination / embryotransfer for 4 weeks

SECONDARY OUTCOMES:
Questionnaire: Intervention rating | 5 minutes before and 5 minutes after insemination / embryotransfer

CONTACTS AND LOCATIONS:
Overall Officials: Joscha Reinhard, Priv-Doz. Dr. med. MBBS BSc, Principal Investigator — Goethe University
Locations (1):
- Klinik für Frauenheilkunde und Geburtshilfe, Frankfurt am Main, Hesse, Germany